CLINICAL TRIAL: NCT02433275
Title: CHildhood ASthma and Environment Research Study - CHASER Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Stefania La Grutta, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Other Study IDs: 8/2014
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
"CHildhood ASthma and Environment Research study - CHASER study" is an observational longitudinal study in outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.

The first phase - transversal study will identify determinants of pediatric asthma control

The second phase - longitudinal study, in patients with persistent asthma, will be focused on:

* predictors for asthma exacerbations and loss of control
* real life adherence to asthma therapy guidelines
* phenotypic characterization through the collection of saliva samples
* assessment of alterations and inflammatory changes in the nasal mucosa through nasal brushing
* evaluation of the presence of 8-isoprostane, nicotine, cotinine and bisphenol-A through urine analysis.

Chaser Project is expected to improve the knowledge of pediatric asthma in patients with different level of control, identifying predictors for asthma exacerbations and loss of control.

ELIGIBILITY:
Inclusion Criteria:

* age 5-16 years
* asthma
* not asthma

Exclusion Criteria:

* chest deformity
* active smoking

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2011-09; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Asthma | 5 years

SECONDARY OUTCOMES:
Measures from saliva samples | 5 years
Measures from nasal brushing | 5 years
Measures from urine samples | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology, IBIM, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
The IPD collected will be available on December 2020.

REFERENCES:
- [Derived] Cilluffo G, Ferrante G, Fasola S, Malizia V, Montalbano L, Ranzi A, Badaloni C, Viegi G, La Grutta S. Association between Asthma Control and Exposure to Greenness and Other Outdoor and Indoor Environmental Factors: A Longitudinal Study on a Cohort of Asthmatic Children. Int J Environ Res Public Health. 2022 Jan 4;19(1):512. doi: 10.3390/ijerph19010512. PMID 35010773
- [Derived] Erkkola RA, Virta LJ, Vahlberg T, Jartti T. Prednisolone for the first rhinovirus induced wheezing reduces use of respiratory medication. Pediatr Allergy Immunol. 2022 Jan;33(1):e13668. doi: 10.1111/pai.13668. Epub 2021 Sep 29. No abstract available. PMID 34536305
- [Derived] Cilluffo G, Han YY, Ferrante G, Dello Russo M, Lauria F, Fasola S, Montalbano L, Malizia V, Forno E, La Grutta S. The Dietary Inflammatory Index and asthma burden in children: A latent class analysis. Pediatr Allergy Immunol. 2022 Jan;33(1):e13667. doi: 10.1111/pai.13667. Epub 2021 Sep 27. PMID 34528308